CLINICAL TRIAL: NCT04234659
Title: Observational Study for Outcomes for Participants With Cardiogenic Shock and Peripartum Cardiomyopathy
Brief Title: PPCM Observational Study (Peripartum Cardiomyopathy)
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Medical College of Wisconsin (Other)
Collaborators: Abiomed Inc. (Industry); University of Pennsylvania (Other)
Responsible Party: Principal Investigator, Sarah Thordsen, Assistant Professor Cardiovascular Medicine, Medical College of Wisconsin
Other Study IDs: PRO35709
Record Dates: First submitted 2019-12-05; First posted 2020-01-21 (Actual); Last update posted 2021-12-13 (Actual); Status verified 2021-12

CONDITIONS: Peripartum Cardiomyopathy; Cardiogenic Shock
MeSH Terms: conditions — Peripartum Cardiomyopathy; Shock, Cardiogenic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Individuals Receiving Mechanical Circulatory Device Support: Individuals receiving mechanical circulatory support device (specifically the IMPELLA® device) for treatment of their index peripartum cardiomyopathy complicated by cardiogenic shock event.
  Interventions: Device: Clinical placement of a temporary IMPELLA® mechanical circulatory support device.
- Individuals Without Mechanical Circulatory Device Support: Individuals not receiving mechanical circulatory support device (specifically the IMPELLA® device) for treatment of their index peripartum cardiomyopathy complicated by cardiogenic shock event.

INTERVENTIONS:
Device: Clinical placement of a temporary IMPELLA® mechanical circulatory support device. — Surgical placement of the IMPELLA® device for life threatening cardiogenic shock not responsive to other medical treatment.
  Groups: Individuals Receiving Mechanical Circulatory Device Support

SUMMARY:
The purpose of this study is to examine the clinical treatment of patients diagnosed with peripartum cardiomyopathy complicated by cardiogenic shock.

DETAILED DESCRIPTION:
This single-site, virtual, longitudinal, observational study will investigate two cohorts (study groups) by enrolling a total of ten participants, five in each cohort. The two cohorts include individuals who received mechanical circulatory support (specifically the IMPELLA® device) compared to individuals who did not receive mechanical circulatory support for treatment of their PPCM complicated by cardiogenic shock index event.

The duration of enrollment for each participant is about 5 months. It is anticipated that the trial will be complete in 12 months. Participant engagement to the study will be self-initiated.

Under the guidance and support of Medical College of Wisconsin research coordinator, participants will directly access the study REDCapTM database for enrollment and follow-up data entry for this study. The research coordinator will obtain and abstract participant medical records documenting the event.

ELIGIBILITY:
Inclusion Criteria:

Females:

* age ≥ 18 years old at the time of entry into the study
* who have capacity to provide consent for study participation
* with self-reported PPCM complicated by cardiogenic shock
* individuals should have US citizenship
* index event occurring within the continental United States.

Exclusion Criteria:

* lack of medical records supporting pregnancy, peripartum cardiomyopathy or cardiogenic shock by study definition
* inability of participant to provide informed consent

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Females meeting study eligibility criteria who have been diagnosed and treated clinically for peripartum cardiomyopathy complicated by cardiogenic shock. A total of 10 participants will be enrolled in each of the two study cohorts (groups).
Sampling Method: Non-Probability Sample
Enrollment: 10 (Estimated)
Dates: Start 2021-01-11 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2023-02-01 (Estimated)

PRIMARY OUTCOMES:
Description of the Long-term Clinical Course of Patients with Peripartum Cardiomyopathy complicated by cardiogenic shock. | From onset of event through 90 days after participant enrollment.
  The retrospective and prospective data collected from study participants will report clinical treatments required to treat the diagnosis of peripartum cardiomyopathy complicated by cardiogenic shock.

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Thordsen, MD, Principal Investigator — Medical College of Wisconsin
Locations (1):
- Medical College of Wisconsin, Milwaukee, Wisconsin, United States

REFERENCES:
- [Background] McNamara DM, Elkayam U, Alharethi R, Damp J, Hsich E, Ewald G, Modi K, Alexis JD, Ramani GV, Semigran MJ, Haythe J, Markham DW, Marek J, Gorcsan J 3rd, Wu WC, Lin Y, Halder I, Pisarcik J, Cooper LT, Fett JD; IPAC Investigators. Clinical Outcomes for Peripartum Cardiomyopathy in North America: Results of the IPAC Study (Investigations of Pregnancy-Associated Cardiomyopathy). J Am Coll Cardiol. 2015 Aug 25;66(8):905-14. doi: 10.1016/j.jacc.2015.06.1309. PMID 26293760
- [Background] Kolte D, Khera S, Aronow WS, Palaniswamy C, Mujib M, Ahn C, Jain D, Gass A, Ahmed A, Panza JA, Fonarow GC. Temporal trends in incidence and outcomes of peripartum cardiomyopathy in the United States: a nationwide population-based study. J Am Heart Assoc. 2014 Jun 4;3(3):e001056. doi: 10.1161/JAHA.114.001056. PMID 24901108
- [Background] Doerr M, Grayson S, Moore S, Suver C, Wilbanks J, Wagner J. Implementing a universal informed consent process for the All of Us Research Program. Pac Symp Biocomput. 2019;24:427-438. PMID 30963079